CLINICAL TRIAL: NCT00697242
Title: Study to Compare the Immunogenicity, Safety and Reactogenicity of GSK Biologicals' (Previously SmithKline Beecham Biologicals') Recombinant Hepatitis B Vaccines With and Without Adjuvant in Healthy Older Adult Volunteers
Brief Title: Comparison of Immuno, Reacto and Safety of Recombinant Hepatitis B Vaccine With or Without MPL in Healthy Older Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 208129/009
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2008-06

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; Engerix™-B; Recombinant Hepatitis B vaccine
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (5):
- Group A (Experimental)
  Interventions: Biological: Recombinant HBsAg with different concentrations of Aluminium Salts and/or MPL
- Group B (Experimental)
  Interventions: Biological: Recombinant HBsAg with different concentrations of Aluminium Salts and/or MPL
- Group C (Experimental)
  Interventions: Biological: Recombinant HBsAg with different concentrations of Aluminium Salts and/or MPL
- Group D (Active Comparator)
  Interventions: Biological: Engerix™-B
- Group E (Experimental)
  Interventions: Biological: Recombinant HBsAg with different concentrations of Aluminium Salts and/or MPL

INTERVENTIONS:
Biological: Engerix™-B — Intramuscular injection, 3 doses
  Arms: Group D
Biological: Recombinant HBsAg with different concentrations of Aluminium Salts and/or MPL — Intramuscular injection, 3 doses
  Arms: Group A; Group B; Group C; Group E

SUMMARY:
In the present study the immunogenicity, reactogenicity and safety of recombinant hepatitis B vaccines with and without MPL will be evaluated in older healthy subjects

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between 50 and 70 years old.
* Written informed consent will have been obtained from the subjects.
* Good physical condition as established by physical examination and history taking at the time of entry

Exclusion Criteria:

* Positive titres for anti hepatitis antibodies
* Any vaccination against hepatitis B in the past.
* Any previous administration of MPL
* Elevated serum liver enzymes at two subsequent determinations 14 days apart.
* History of significant and persisting hematologic, hepatic, renal, cardiac or respiratory disease.
* Axillary temperature > 37.5°C at the time of injection.
* Any acute disease at the moment of entry.
* Chronic alcohol consumption.
* Any treatment with immunosuppressive or immunostimulant therapy.
* Any chronic drug treatment, which in the investigator's opinion, precludes inclusion into the study.
* History of allergic disease likely to be stimulated by any component of the vaccine.
* Administration of any other vaccine(s) or any immunoglobulin during the study period.
* Simultaneous participation in any other clinical trial.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 1994-01; Primary Completion 1995-11 (Actual); Study Completion 1995-11 (Actual)

PRIMARY OUTCOMES:
Anti-hepatitis B surface antigen (HBs) antibody concentrations | At M2 and M7

SECONDARY OUTCOMES:
Anti-pre-S1 antibody concentrations | Screening, Months 1, 2, 3, 6, 7, 8 and 12, depending on group allocation
Anti-HBs antibody concentrations | Screening, Months 1, 2, 3, 6, 7, 8 and 12
Occurrence and intensity of local and general solicited symptoms | 4-day after vaccination
Cell mediated immunity | Month 0, Month 2 and month 7
Occurrence of unsolicited adverse events | 30 days after vaccination
Occurrence of serious adverse events | During the study period and 30 days after last vaccine dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Clinical Trials Call Center, Vienna, Austria
- GSK Clinical Trials Call Center, Ghent, Belgium
- GSK Clinical Trials Call Center, Hvidovre, Denmark
- GSK Clinical Trials Call Center, Reykjavik, Iceland